CLINICAL TRIAL: NCT04117230
Title: Clinical Outcomes in Patients in Need of a Non-permanent Extracorporeal Cardiocirculatory Support System (Peripheral Extracorporeal Membrane Oxygenation (ECMO) or Axial Flow Pump IMPELLA)
Brief Title: CARDSUP - SWISS Circulatory Support Registry
Acronym: CARDSUP
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 4075
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project's main goal is to collect baseline clinical and procedural data as well as to assess clinical outcomes for all patients undergoing ECMO or Impella implantation at all included sites. All patients undergoing ECMO and/or IMPELLA implantation will be prospectively registered. Device use is according to the decision of the treating physician and independent of this registry.

DETAILED DESCRIPTION:
This prospective data collection is made up of an all-comers design, including all eligible consecutive patients receiving an Impella (2.5, 5, CP, or RP) or VA-ECMO device via femoral access who gave their consent (or, if not possible, their relative).

The project's main goal is to collect baseline clinical and procedural data as well as to assess clinical outcomes for all patients undergoing ECMO or Impella implantation at all included sites. All patients undergoing ECMO and/or IMPELLA implantation will be prospectively registered. Device use is according to the decision of the treating physician and independent of this registry.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Medical indication for implantation of a peripheral cannulated VA-ECMO or microaxial flow pump (IMPELLA) or newer LV / LA-Ascending Aorta devices.
* Signed informed consent by patient or relative or waived consent by EC

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In an all-comers design, every patient receiving an MCS will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-08-09 (Actual); Primary Completion 2034-08-31 (Estimated); Study Completion 2034-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of deceased participants at 1 month after cardiogenic shock | 30 days
  All-cause mortality at 30 days

SECONDARY OUTCOMES:
Statistical and medical analysis of major adverse cardiac and cerebrovascular events (MACCE) reported by participants | 6 months
  Major adverse cardiac and cerebrovascular events (MACCE)
Statistical and medical analysis of vascular complications (VARC) reported by participants | 6 months
  Vascular complications (VARC)
Statistical and medical analysis of vascular surgery needed by participants | 6 months
  Need for vascular surgery
Statistical and medical analysis of bleeding complications (minor, major) reported by participants | 6 months
  Bleeding complications (minor, major)
Implantation time of MCS-device | 6 months
  Implantation time of MCS-device
Support time under MCS | 6 months
  Support time under MCS
Analysis of New York Heart Association (NYHA) Classification for participants | 6 months
  The New York Heart Association (NYHA) Classification provides a way of classifying the extent of heart failure. It classifies patients in one of four categories based on their limitations during physical activity; the limitations/symptoms are in regards to normal breathing and varying degrees in shortness of breath and or angina pain. Class I is defined as no symptoms and no limitation in ordinary physical activity worsening to Class IV defined as severe limitations.
Modified rankin scale | 6 months
  Modified rankin scale measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological Disability. The scale ranges form 0-6 with 0 defined as no Symptoms and 5 being severe Symptoms and 6 defined as death.
Number of deceased participants at 6 month after cardiogenic shock | 6 months
  Mortality at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lukas C Hunziker Munsch, Prof MD, Study Chair — University of Bern
Locations (5):
- Switzerland (5):
  - Universitätsspital Basel, Basel
  - Insel Gruppe AG, Inselspital Bern, Bern
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital Winterthur, Winterthur
  - Stadtspital Treimli, Zurich